CLINICAL TRIAL: NCT03913754
Title: Psychosocial Consequences of Systemic Lupus Erythematosus: a Study of Patients and Their Spouses Psy-LUP Study
Brief Title: Psycho-social Consequences of Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-29
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lupus Erythematosus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lupus Patients with kidneys failure: Assessment of quality of life on everydays life trough questionnare
  Interventions: Other: Psycho-social consequences of lupus erythematosus
- Lupus Patients without kidneys failure: Assessment of quality of life on everydays life trough questionnare
  Interventions: Other: Psycho-social consequences of lupus erythematosus

INTERVENTIONS:
Other: Psycho-social consequences of lupus erythematosus — It will be necessary to take into account the psychosocial experience of the disease [47] and to allow a narrative exploration of this experience and its psycho-social consequences both for the patients and their spouses (ie the experiential dimension of the disease in connection with the life trajectory, the life of a couple, elaborate representations concerning the disease). The purpose of this approach is not only to question the meaning of the disease (beliefs, representations), the psycho-social management of the disease, its inclusion in the socio-cultural condition of the patients, but also to allow an analysis of the inscription. of the disease in the relationship and its implications (relational, affective, sexual) and its impact on the possibilities of social participation.

SUMMARY:
this project will allow us to evaluate and understand the impact of SLE on the couple's life and its relational and affective components. In addition, the Psy-LUP study will describe the representations that sick people and their relatives have of lupus disease. All the data collected will make it possible to target interventions with 1) patients and their relatives, in terms of therapeutic education, psychosocial support, support groups (associations); 2) caregivers caring for people with SLE, so that they can integrate the issues of the patient's experience in their care practice and their reflection on therapeutic strategies.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a rare chronic autoimmune disease (1/2000 inhabitants) that evolves in periods of recurrent remissions. Sufferers are most often young women of childbearing age. SLE affects the life of a couple like family life (financial, emotional, relational or sexual conditions of the couple). In addition, the disease and its treatments can hinder the possibility of building a family project (pregnancy).

The purpose of the Psy-LUP study is to study the impact of SLE on the social participation of patients, that is to say on their ability to get involved in different areas of daily life. These repercussions could be all the more important as lupus disease is active and complicated by severe diseases such as kidney disease. We want to study how sick people and their loved ones (spouse in particular) think about lupus disease, how it fits into their life history, how people have adapted to this disease, and how it affects their lives. could have on their social participation, their social support, their life of couple. The Psy-LUP study will be carried out in different care services, and by telephone interviews at home, with two main axes: (1) a study by questionnaire with patients (n = 100); (2) a qualitative study through research interviews with patients (n = 40) and their spouses (n = 20). The realization of this project will allow us to evaluate and understand the impact of SLE on the life of the couple and its relational and affective components. In addition, the Psy-LUP study will describe the representations that sick people and their relatives have of lupus disease. All the data collected will make it possible to target interventions with 1) patients and their relatives, in terms of therapeutic education, psychosocial support, support groups (associations); 2) caregivers caring for people with SLE, so that they can integrate the issues of the patient's experience in their care practice and their reflection on therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Presenting an LES according to ACR or SLICC criteria
* Being followed in Marseille in Nephrology or Internal Medicine as part of the Competence Center Lupus PACA
* Having agreed to participate in the study after information

Exclusion Criteria:

* Minor person
* Person deprived of liberty
* Person not affiliated to a social security scheme

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population covered by the QuaNTi Psy-LUP project is that of patients monitored by the Lupus PACA Competence Center, and a cohort of SLE patients with renal impairment (WIN-Lupus trial).
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
the physical, psychological and social impact of chronic diseases | 12 months
  Quality of life scale Short Study Form-36 (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- Assitance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Background] Aim MA, Queyrel V, Tieulie N, Chiche L, Faraut J, Manet C, Schleinitz N, Harle JR, Jourde-Chiche N, Dany L. Importance of temporality and context in relation to life habit restrictions among patients with systemic lupus erythematosus: A psychosocial qualitative study. Lupus. 2022 Oct;31(12):1423-1433. doi: 10.1177/09612033221115966. Epub 2022 Aug 2. PMID 35916586
- [Background] Manet C, Aim MA, Queyrel V, Faraut J, Costedoat-Chalumeau N, Daugas E, Hachulla E, Harle JR, Huart A, Hummel A, Kaplanski G, Mazodier K, Mancini J, Sarrot-Reynauld F, Schleinitz N, Swiader L, Tieulie N, Manet P, Dany L, Chiche L, Jourde-Chiche N. Determinants of social participation in patients living with systemic lupus erythematosus: the Psy-LUP multicentre study. RMD Open. 2025 Jun 25;11(2):e005661. doi: 10.1136/rmdopen-2025-005661. PMID 40562684